CLINICAL TRIAL: NCT01355406
Title: Evaluation of Safety and Efficacy of the FlexStent® Femoropopliteal Self-Expanding Stent System Study
Brief Title: Evaluation of Safety and Efficacy of the FlexStent® Femoropopliteal Self-Expanding Stent System
Acronym: OPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Massachusetts General Hospital (Other); Prairie Education and Research Cooperative (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSS-0003
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Vascular Disease; Cardiovascular Diseases; PAD
Keywords: FlexStent; Superficial Femoral Artery or SFA; Self Expanding Stent; Stent; Bare Metal Stent
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAD (Other): This is a prospective single-arm multi-center clinical trial designed to evaluate the safety and efficacy of the Flexible Stenting Solutions Flext Stent® Femoropopliteal stenting system in subjects with lower limb peripheral arterial desease (PAD). Subjects targeted for enrollment must have a single de-novo lesion located in the superficial femoral artery and/or proximal popliteal artery with at > 70% stenosis. Subjects must meet all enrollment criteria and provide written informed consent prior to participation in the study.
  Interventions: Device: FlexStent® Femoropopliteal Self Expanding Stent System

INTERVENTIONS:
Device: FlexStent® Femoropopliteal Self Expanding Stent System — Transcatheter over guidewire placement of an intravascular stent(s)
  Other Names: FlexStent®; OPEN

SUMMARY:
This is a clinical study of a new self-expanding stent (FlexStent®) designed specifically to cope with the extreme demands of the superficial femoral artery (SFA)/proximal popliteal artery. The arteries are often abbreviated as femoropopliteal.

The intent of this study is to demonstrate that the FlexStent® Femoropopliteal Self-Expanding Stent System is safe and effective for the treatment of patients with peripheral arterial disease. Specifically, the FlexStent® shall meet or exceed the proposed safety and efficacy performance goals established for Femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria:

1. Subjects, male or female, must be at least 35 years of age at the time of consent. A female of childbearing potential may be enrolled, provided she has a negative pregnancy test within 7 days of screening.
2. Subjects must give written informed consent prior to participation in the study and must understand the purpose of this study and be willing to adhere to the study procedures described in this protocol.
3. Rutherford Classification Category 2-4
4. De novo lesion in the Femoropopliteal artery, including the entire extent of the superficial femoral artery and the proximal portion of the popliteal artery extending to the medial condyle 3 cm above the knee joint
5. Disease segment length ≤ 180 mm
6. >70% diameter stenosis and/or occlusion based on site-determined visual angiography
7. Patent ipsilateral iliac artery
8. Patency of ipsilateral mid/distal popliteal artery and at least 1 tibial artery with no planned intervention
9. Target reference vessel diameter 3.5-7.5 mm.
10. Projected life expectancy of 12 months or greater
11. Patient is available for follow-up for 36 months and is willing and able to comply with all follow-up requirements
12. Patient is willing and able to provide signed informed consent

Exclusion Criteria:

Any subject meeting any of the following criteria will be excluded from the study.

1. Target vessel previously treated with a stent
2. Target lesion within 1.5 cm of the ostium of the SFA
3. Rutherford Classification Category 0,1,5 or 6
4. Inability to tolerate antithrombotic or antiplatelet therapies
5. Pregnancy (female of child-bearing age confirmed pregnant)
6. Other comorbidity risks which in the opinion of the investigator limit longevity or likelihood of complying with protocol follow up.
7. Serum creatinine > 2.5 mg/dL
8. Myocardial infarction or stroke within 30 days of treatment date
9. Known hypercoagulable state
10. Known bleeding diathesis
11. Untreated angiographically-evident thrombus in target vessel
12. Patients currently enrolled in any other clinical trial

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is freedom from all cause death, TLR, or index limb amputation through 30 days. | 30 Days
  The primary safety endpoint is defined as freedom from all cause death, index limb amputation and target lesion revascularization (TLR) through 30 days. The proportion of patients remaining free from this composite endpoint will be compared to a safety performance goal for bare nitinol stents.
The primary efficacy endpoint is vessel patency at 12 months. | 12 Months
  The primary efficacy endpoint is vessel patency at 12 months. Vessel patency is defined as freedom from a greater than 50% restenosis in the stented segment as determined by the DUS peak systolic velocity ratio (PSVR) comparing data within the treated segment to the proximal normal arterial segment and freedom from clinically-driven TLR within the stented segment within 1 year of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: William A. Gray, MD, Principal Investigator — Center for Interventional Vascular Therapy / Columbia University Medical Center
Locations (38):
- United States (36):
  - Abrazo Health Care Clinical & Trans. Research, Phoenix, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - El Camino Hospital, Mountain View, California
  - Yale University/New Haven Hospital, New Haven, Connecticut
  - Manatee Memorial Hospital, Bradenton, Florida
  - Florida Research Network, Gainesville, Florida
  - Memorial Hospital, Jacksonville, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Mount Sinai Miami Medical Center, Miami Beach, Florida
  - Florida Hospital Pepin Heart Institute, Tampa, Florida
  - University Hospital, Augusta, Georgia
  - St. John's Hospital, Springfield, Illinois
  - Midwest Cardiovascular Research Foundation / Trinity Medical Center, Davenport, Iowa
  - Healient Physician Group, Overland Park, Kansas
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Christus St. Patrick Hospital, Lake Charles, Louisiana
  - Glenwood Regional Medical Center, West Monroe, Louisiana
  - Washington Adventist Hospital / Center for Cardiac & Vascular Research, Takoma Park, Maryland
  - Deborah Heart, Browns Mills, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Our Lady of Lourdes Medical Center, Haddon Heights, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Gotham Cardiovascular Research, PC, New York, New York
  - Columbia University Medical Center, Center for Interventional Vascular Therapy, New York, New York
  - CarolinaEast Health Center, New Bern, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Sanford Research/USD/Sanford Clinic, Fargo, North Dakota
  - Riverside Methodist Hospital / MidWest Cardiology Research Foundation, Columbus, Ohio
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Allegheny General Hospital/Forbes Hospital, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Providence Sacred Heart Medical Center / Providence Spokane Cardiology, Spokane, Washington
  - Wisconsin Heart Hospital, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center / Aurora Medical Group, Milwaukee, Wisconsin
- Belgium (2):
  - Imelda Hospital / Flanders Medical Research Program, Bonheiden
  - A.Z. Sint-Blasius Hospital / Flanders Medical Research Program, Dendermonde

REFERENCES:
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972